CLINICAL TRIAL: NCT04084210
Title: Understanding the Real-World Impact of the Use of Three Alternate Nicotine-Delivery Products on Combustible Cigarette Use
Brief Title: Impact of Alternative Nicotine-Delivery Products on Combustible Cigarette Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2019-0252; 1R01CA239309 (NIH); A534253 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*G (Other: UW Madison); Protocol Version 2/17/2021 (Other: UW Madison)
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: For this mixed design study, 180 daily adult smokers who are not planning to quit smoking will be randomly assigned to one of three levels of the between-subjects factor: 1) VLNCs; 2) Juul e-cigarettes; or 3) no alternative product. During two different weeks, participants will be asked to switch from their usual cigarettes and use only study products. They will also be asked to use either an active nicotine or placebo patch (the within-subjects factor), provided in double-blind fashion and counterbalanced order.
  It should be noted that there were no significant within-subject effects (i.e. comparing Juul + Active Patch in Wk 1 and Placebo Patch in Wk 2 vs. JUUL + Placebo Patch in Wk 1 then Active Patch in Wk 2 yielded no significant differences) therefore results are presented as a 3-group parallel design (i.e. Juul + Active vs. Placebo Patch, VLNC + Active vs. Placebo Patch, No Product + Active vs. Placebo Patch).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned to Juul, Very Low Nicotine Cigarette, or No Product with no masking of product type. However, participants will be randomly assigned to receive either placebo or active nicotine patch with masking regarding placebo vs active patch.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Juul + Active Patch in Wk 1 and Placebo Patch in Wk 2 (Active Comparator): Participants will be given Juul e-cigarettes for four weeks; in Switch Week 1, participants also will use active nicotine patches; in Switch Week 2, participants will use placebo patches.
  Interventions: Device: Juul Electronic cigarette; Drug: Active Nicotine Patch; Other: Placebo Patch
- Juul + Placebo Patch in Wk 1 and Active Patch in Wk 2 (Active Comparator): Participants will be given Juul e-cigarettes for four weeks; in Switch Week 1, participants also will use placebo patches; in Switch Week 2, participants will use active nicotine patches.
  Interventions: Device: Juul Electronic cigarette; Drug: Active Nicotine Patch; Other: Placebo Patch
- VLNC + Active Patch in Wk 1 and Placebo Patch in Wk 2 (Active Comparator): Participants will be given very low nicotine cigarettes (VLNCs) for four weeks; in Switch Week 1, participants also will use active nicotine patches; in Switch Week 2, participants will use placebo patches.
  Interventions: Other: Very Low Nicotine Cigarettes; Drug: Active Nicotine Patch; Other: Placebo Patch
- VLNC + Placebo Patch in Wk 1 and Active Patch in Wk 2 (Active Comparator): Participants will be given very low nicotine cigarettes (VLNCs) for four weeks; in Switch Week 1, participants also will use placebo patches; in Switch Week 2, participants will use active nicotine patches.
  Interventions: Other: Very Low Nicotine Cigarettes; Drug: Active Nicotine Patch; Other: Placebo Patch
- No Product + Active Patch in Wk 1 and Placebo Patch in Wk 2 (Other): Participants will be given no alternative nicotine delivery products but in Switch Week 1, participants will use active nicotine patches; in Switch Week 2, participants will use placebo patches.
  Interventions: Drug: Active Nicotine Patch; Other: Placebo Patch
- No Product + Placebo Patch in Wk 1 and Active Patch in Wk 2 (Other): Participants will be given no alternative nicotine delivery products for two weeks but in Switch Week 1 participants will use placebo patches; in Switch Week 2, participants will use active nicotine patches.
  Interventions: Drug: Active Nicotine Patch; Other: Placebo Patch

INTERVENTIONS:
Device: Juul Electronic cigarette — The juul e-cigarette pods contain 0.7 ml nicotine by volume / 5% nicotine by weight.
  Other Names: Juul
  Arms: Juul + Active Patch in Wk 1 and Placebo Patch in Wk 2; Juul + Placebo Patch in Wk 1 and Active Patch in Wk 2
Other: Very Low Nicotine Cigarettes — These very low nicotine cigarettes (VLNCs) consist of reduced nicotine cigarettes containing 0.03 mg of nicotine; these VLNCs were obtained from National Institute on Drug Abuse (NIDA's) Drug Supply Program (NOT-DA-14-004).
  Other Names: VLNC
  Arms: VLNC + Active Patch in Wk 1 and Placebo Patch in Wk 2; VLNC + Placebo Patch in Wk 1 and Active Patch in Wk 2
Drug: Active Nicotine Patch — Active nicotine patches, with dosing based on the package insert (>10 cigs/day = 21 mg patch and <11 cigs/day = 14 mg patches).
  Other Names: Nicotine Patch
Other: Placebo Patch — Placebo patch containing no nicotine.

SUMMARY:
The goal of this research is to understand the potential impact of two new FDA strategies to ensure the availability of safer Alternative Nicotine Delivery Systems (ANDS) and to reduce the nicotine content in combustible cigarettes to non-addictive levels. Specifically, this research will examine how well ANDS and very low nicotine cigarettes (VLNCs) can work alone or in combination with the current strategy of providing a safe source of nicotine via nicotine replacement medications to reduce use of combustible cigarettes, in real-world settings.

The investigators will enroll 180 daily adult smokers who are not planning to quit smoking within the next 30 days into this mixed design study. Participants will be randomly assigned to one of three levels of the between-subjects factor: 1) VLNC cigarettes; 2) Juul e-cigarettes (with nicotine); or 3) no alternative product. Participants receiving an alternative product (VLNC or e-cigarettes) will be asked to use it for 4 weeks (Weeks 1 through 4). During Weeks 2 and 4 all participants will be asked to switch from their cigarettes to use only study products (i.e., Juul e-cigarettes, VLNCs, or no alternative product) and to use either an active nicotine or placebo patch (the within-subjects factor), provided in double-blind fashion and counterbalanced order. During Weeks 1 through 4, participants will use a smartphone to record, in the moment, each time they use their own cigarettes or any alternative product. For a random daily subset of use events, participants will complete additional questions about the internal and external context of their use (e.g., affect, any restrictions on smoking) and their response to use (e.g., withdrawal alleviation, taste, satisfaction). Using these data, the investigators will also examine the effects of these products on the rewarding value of smoking and possible mechanisms driving such behavior (e.g., withdrawal alleviation, satisfaction, taste).

This research will provide critical information regarding the potential impact of providing cigarettes with non-addictive levels of nicotine and safe ANDS, with or without nicotine replacement, in real-world settings on smokers' use of their usual cigarettes and other outcomes. Information on the short-term effects of products that could be accessible in the future will provide data that could inform regulatory policy decisions regarding the public health impact of safe ANDS and non-addictive cigarettes.

DETAILED DESCRIPTION:
Design and Objective: The primary goal of this research is to assess the ability of alternative products (VLNCs vs. e-cigs vs. no alternative product; between-subjects factor) to serve as a substitute for conventional cigarettes and how this is influenced by steady-state nicotine (nicotine vs. placebo patches; within-subjects factor). In addition, the investigators will explore the contexts in which participants are and are not able to switch from their conventional cigarettes. Such contextual information will provide insight into internal (i.e., withdrawal, expectancies) and external environments (i.e., being around smokers, smoking restrictions) that promote or interfere with switching behavior. The investigators will also explore person factors and beliefs that may drive alternative product use and substitution success. Person factors that may influence use behavior include sex (a key biological variable), education level, dependence, instrumental smoking motives (e.g., smoking for affect regulation, taste, or social experiences), and psychiatric comorbidity. Beliefs that may influence use behavior include beliefs about the safety and addiction potential of conventional cigarettes and the alternative products. Understanding the relation of person factors and beliefs with use behavior could inform regulatory actions related to product labeling and education. Finally, the investigators will explore potential mechanisms that might drive use behavior and support substitution.

This research will enroll 180 adult smokers in a mixed design study with a within-subjects factor (active nicotine patch vs. placebo patch) and a between-subjects factor (alternative products: VLNCs, e-cigs, or no product). Participants will be randomized to receive either 4 weeks of VLNCs, 4 weeks of e-cigs, or no alternative product. After one week practicing with the alternative product, participants will complete the first of two 7-day switching trials during which they will be asked to refrain from smoking their own cigarettes and encouraged to use the alternative product to which they have been assigned (although the no alternative product group will not have any other products to use). All participants will be given patches (active nicotine or placebo, in counterbalanced order) to use during the Switch Week. After this first Switch Week, participants will smoke normally for one week and then have their second Switch Week using the other type of patch (active or placebo). Participants will complete Ecological Momentary Assessments (EMAs) on smartphones at baseline and during the 4 weeks of product use. EMA targets include own cigarette use, alternative product use, withdrawal symptoms, rewarding value of product use (e.g., taste, buzz), and environmental and affective context of any tobacco product use. The investigators will then conduct a 3-month follow-up to assess cigarette and e-cig use, risk perceptions, and future use intentions.

This design addresses the six critical methodological issues for understanding the impact of alternative products outlined by Villanti et al.: 1) rigorous assessment of the key outcome (conventional cigarettes smoked); 2) assessment of product use during switching; 3) use of appropriate control/comparison groups; 4) measurement of product exposure/use that precedes switching; 5) evaluation of the dose and duration of product exposure/use; and 6) clear evaluation of the type and quality of the products used (e.g., satisfaction).

Recruitment and Participants: Participants from the greater Madison and Milwaukee, Wisconsin areas will be recruited via media recruitment methods (i.e., television, newspaper, and earned media) that have recruited thousands of smokers. Investigators will also use Internet/Facebook advertisements that have been successful in recent e-cig studies that recruited 422 smokers willing to provide EMA data during seven 2-week assessment periods over 2 years and 74 dual users willing to reduce combustible cigarette use and switch to using only e-cigs. Given this, it is feasible to recruit 180 smokers for this study within 18 months.

Procedures and Measures: Interested smokers will complete a phone screen to determine initial eligibility. Potentially eligible smokers will attend an orientation visit where, after providing a breath sample to verify eligibility (CO > 6 ppm), they will receive a detailed description of the study and provide written informed consent, and complete baseline assessments. At Visit 1, participants will be randomized to receive VLNCs, e-cigs, or no alternative product and will be trained to use the product. The study database will randomize participants, stratified by clinic, gender, and race [White vs. Non-White], to enhance scientific rigor and reproducibility. Participants will be trained to use the smartphone to complete daily assessments, using the training that was effective in prior research, and will schedule future study visits. Participants will use their alternative products as they would like for one week to become comfortable with the product. At Visit 2, participants will complete assessments, provide a breath sample for CO assessment and a urine sample for cotinine assessment, receive feedback on their compliance with the smartphone assessments, and be given study patches to use during Switch Week 1 when they will be asked to abstain from using their own cigarettes for the week. Participants will then attend a mid-Switch Week visit (Visit 3) and an end-of-Switch Week visit (Visit 4) to assess biomarkers (a breath sample for CO assessment and a urine sample for cotinine). At Visit 4, the end of Switch Week 1, participants will be told that they can smoke as usual for a week. Then, at the start of Switch Week 2 (Visit 5), participants will be given the other type of patch (active or placebo) and asked to abstain from smoking their own cigarettes for a week. As during the prior Switch Week, participants will attend visits mid-week and at the end of the week to assess biomarkers (Visits 6 and 7). The investigators will attempt to schedule appointments at the same time of day (i.e., within a 2-hour window) for each participant so that there is consistent time for product use prior to providing the biological samples across study visits. Participants will complete a follow-up assessment call at 3 months. The baseline visit will last 2 hours, but subsequent visits will last <30 minutes. Participants will carry a smartphone to complete EMAs from Orientation through all 4 weeks of product use.

Knowledge to be Gained: The results from this research will provide important insight into how well very low nicotine cigarettes and e-cigarettes serve as a substitute for conventional cigarettes and how this is influenced by the presence of steady-state nicotine. Further, these data will inform scientists and regulators about the potential mechanisms that may support the use of alternative products. This information will aid scientists and regulatory bodies in understanding the real-world impact of potential regulatory policies regarding access to safer nicotine sources and reducing the addiction potential of combustible tobacco products.

ELIGIBILITY:
Inclusion criteria:

* smoking >4 cigarettes/day for the previous 6 months
* able to read, write, and speak English
* no plans to quit smoking in the next 30 days
* not currently taking smoking cessation medication
* willing and medically able to use nicotine patches
* exhaled carbon monoxide (CO) > 6 ppm.

Exclusion criteria:

* currently in treatment for psychosis or bipolar disorder
* e-cigarette use within the last month
* currently pregnant or breastfeeding.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Piper, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin Center for Tobacco Research and Intervention, Madison, Wisconsin
  - UW Center for Tobacco Research and Intervention, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
We will make the set of final de-identified datasets available in encrypted standard file formats or secure File Transfer Protocol (FTP) transmission by request from other researchers in a timely manner (no later than the acceptance for publication of the main findings from the final dataset).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the publication of the main findings
Access Criteria: Approval of a data request by the investigators

REFERENCES:
- [Derived] Piper ME, Kaye JT, Piasecki TM, Yang JJ, Buu A. Cannabis use among adults who smoke tobacco: Relations with switching from combusted cigarettes to e-cigarettes or very low nicotine cigarettes. Drug Alcohol Depend. 2025 Oct 1;275:112821. doi: 10.1016/j.drugalcdep.2025.112821. Epub 2025 Aug 6. PMID 40803048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from the greater Madison and Milwaukee, WI areas were recruited via media recruitment methods (i.e., TV, newspaper, and earned media) and paid Facebook advertisements. Of the 2036 potential participants, 209 (10.3%) were eligible, provided consent and were randomized. Of those randomized, 160 completed both switch weeks and were included in the analyses.
Groups:
- Juul + Active Patch in Wk 1 and Placebo Patch in Wk 2: Participants will be given Juul e-cigarettes for four weeks; in Switch Week 1 - half of participants will use active nicotine patches and half will use placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 will use placebo patches, and the participants who received placebo patches during Switch Week 1 will use active nicotine patches.
  Juul Electronic cigarette: The juul e-cigarette pods contain 0.7 ml nicotine by volume / 5% nicotine by weight.
  Active Nicotine Patch: Active nicotine patches, with dosing based on the package insert (>10 cigs/day = 21 mg patch and <11 cigs/day = 14 mg patches).
  Placebo Patch: Placebo patch containing no nicotine.
- VLNC + Active Patch in Wk 1 and Placebo Patch in Wk 2: Participants will be given very low nicotine cigarettes (VLNCs) for four weeks; in Switch Week 1 - half of participants will use active nicotine patches and half will use placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 will use placebo patches, and the participants who received placebo patches during Switch Week 1 will use active nicotine patches.
  Very Low Nicotine Cigarettes: These very low nicotine cigarettes (VLNCs) consist of reduced nicotine cigarettes containing 0.03 mg of nicotine; these VLNCs were obtained from National Institute on Drug Abuse (NIDA's) Drug Supply Program (NOT-DA-14-004).
  Active Nicotine Patch: Active nicotine patches, with dosing based on the package insert (>10 cigs/day = 21 mg patch and <11 cigs/day = 14 mg patches).
  Placebo Patch: Placebo patch containing no nicotine.
- No Product + Active Patch in Wk 1 and Placebo Patch in Wk 2: Participants will be given no alternative nicotine delivery products but in Switch Week 1 - half of participants will use active nicotine patches and half will use placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 will use placebo patches, and the participants who received placebo patches during Switch Week 1 will use active nicotine patches.
  Active Nicotine Patch: Active nicotine patches, with dosing based on the package insert (>10 cigs/day = 21 mg patch and <11 cigs/day = 14 mg patches).
  Placebo Patch: Placebo patch containing no nicotine.
Period: Overall Study
Arm/Group | Juul + Active Patch in Wk 1 and Placebo Patch in Wk 2 | Juul + Placebo Patch in Wk 1 and Active Patch in Wk 2 | VLNC + Active Patch in Wk 1 and Placebo Patch in Wk 2 | VLNC + Placebo Patch in Wk 1 and Active Patch in Wk 2 | No Product + Active Patch in Wk 1 and Placebo Patch in Wk 2 | No Product + Placebo Patch in Wk 1 and Active Patch in Wk 2
Started | 34 | 32 | 37 | 36 | 34 | 36
Completed | 27 | 27 | 29 | 24 | 26 | 27
Not Completed | 7 | 5 | 8 | 12 | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Juul + Active and Placebo Patch: Participants will be given Juul e-cigarettes for four weeks; in Switch Week 1 - half of participants will use active nicotine patches and half will use placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 will use placebo patches, and the participants who received placebo patches during Switch Week 1 will use active nicotine patches.
  Juul Electronic cigarette: The Juul e-cigarette pods contain 0.7 ml nicotine by volume / 5% nicotine by weight.
  Active Nicotine Patch: Active nicotine patches, with dosing based on the package insert (>10 cigs/day = 21 mg patch and <11 cigs/day = 14 mg patches).
  Placebo Patch: Placebo patch containing no nicotine.
- VLNC + Active and Placebo Patch: Participants will be given very low nicotine cigarettes (VLNCs) for four weeks; in Switch Week 1 - half of participants will use active nicotine patches and half will use placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 will use placebo patches, and the participants who received placebo patches during Switch Week 1 will use active nicotine patches.
  Very Low Nicotine Cigarettes: These very low nicotine cigarettes (VLNCs) consist of reduced nicotine cigarettes containing 0.03 mg of nicotine; these VLNCs were obtained from National Institute on Drug Abuse (NIDA's) Drug Supply Program (NOT-DA-14-004).
  Active Nicotine Patch: Active nicotine patches, with dosing based on the package insert (>10 cigs/day = 21 mg patch and <11 cigs/day = 14 mg patches).
  Placebo Patch: Placebo patch containing no nicotine.
- No Product + Active and Placebo Patch: Participants will be given no alternative nicotine delivery products but in Switch Week 1 - half of participants will use active nicotine patches and half will use placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 will use placebo patches, and the participants who received placebo patches during Switch Week 1 will use active nicotine patches.
  Active Nicotine Patch: Active nicotine patches, with dosing based on the package insert (>10 cigs/day = 21 mg patch and <11 cigs/day = 14 mg patches).
  Placebo Patch: Placebo patch containing no nicotine.
- Total: Total of all reporting groups
Arm/Group | Juul + Active and Placebo Patch | VLNC + Active and Placebo Patch | No Product + Active and Placebo Patch | Total
Number analyzed (Participants) | 54 | 53 | 53 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.37 (9.57) | 52.00 (13.26) | 51.21 (13.22) | 51.86 (12.06)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Transgender | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Population: See added Baseline Measure Sex/Gender Customized for Transgender participant.
  Participants
    number analyzed (Participants) | 53 | 53 | 53 | 159
    Female | 34 | 34 | 28 | 96
    Male | 19 | 19 | 25 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 50 | 48 | 51 | 149
  Unknown or Not Reported | 2 | 3 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 10 | 15 | 35
  White | 40 | 38 | 35 | 113
  More than one race | 4 | 1 | 1 | 6
  Unknown or Not Reported | 0 | 2 | 2 | 4
Cigarettes per day (CPD) [Mean (Standard Deviation); unit: cigarettes per day] | 17.29 (9.89) | 16.78 (9.3) | 17.55 (9.59) | 16.85 (9.34)

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Conventional Cigarettes Smoked During Each Switch Week
Description: The mean number of conventional cigarettes smoked during each Switch Week will be used as a measure for conventional cigarette usage.
Time Frame: During the two 1-week switching periods
Measure: Mean (Standard Deviation); unit: Cigarettes per day
Arm/Group | Juul + Active and Placebo Patch | VLNC + Active and Placebo Patch | No Product + Active and Placebo Patch
Number analyzed (Participants) | 54 | 53 | 53
Cigarettes per day
  Cigarettes per day during Placebo Patch Switch Week | 3.2 (3.6) | 3.2 (4.8) | 5.8 (6.2)
  Cigarettes per day during Active Patch Switch Week | 3.1 (3.3) | 2.9 (4.6) | 5.1 (5.5)

2. Secondary Outcome: Mean Number of VLNCs Smoked or Vape Events Per Day Reported During Each Switch Week
Description: The mean number of VLNCs smoked or vape events reported per day during each Switch Week will be used as a measure of alternative product use.
Time Frame: During the two 1-week switching periods
Measure: Mean (Standard Deviation); unit: events per day
Arm/Group | Juul + Active and Placebo Patch | VLNC + Active and Placebo Patch | No Product + Active and Placebo Patch
Number analyzed (Participants) | 54 | 53 | 53
events per day
  Product Use per day during Placebo Patch Switch Week | 7.46 (4.49) | 10.09 (8.39) | 0.0 (0.0)
  Product Use per day during Active Patch Switch Week | 6.61 (3.82) | 8.64 (6.99) | 0.0 (0.0)

ADVERSE EVENTS:
Time Frame: All participants were assessed for adverse events at all study visits over the course of 4 weeks.
Groups:
- JUUL + Active Patch: Participants were given Juul e-cigarettes for four weeks; in Switch Week 1 - half of participants used active nicotine patches and half used placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 used placebo patches during Switch Week 2, and the participants who received placebo patches during Switch Week 1 used active nicotine patches during Switch Week 2. AEs were assessed during Switch Weeks as well as during times when participants were smoking as usual and/or using JUUL, but not using nicotine patches.
  These data are AEs for subjects during the week that they were using JUUL and Active Patches.
  Juul Electronic cigarette: The Juul e-cigarette pods contain 0.7 ml nicotine by volume / 5% nicotine by weight.
  Active Nicotine Patch: Active nicotine patches, with dosing based on the package insert (>10 cigs/day = 21 mg patch and <11 cigs/day = 14 mg patches).
- JUUL + Placebo Patch: Participants were given Juul e-cigarettes for four weeks; in Switch Week 1 - half of participants used active nicotine patches and half used placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 used placebo patches during Switch Week 2, and the participants who received placebo patches during Switch Week 1 used active nicotine patches during Switch Week 2. AEs were assessed during Switch Weeks as well as during times when participants were smoking as usual and/or using JUUL, but not using nicotine patches.
  These data are AEs for subjects during the week that they were using JUUL and Placebo Patches.
  Juul Electronic cigarette: The Juul e-cigarette pods contain 0.7 ml nicotine by volume / 5% nicotine by weight.
  Placebo Patch: Placebo patch containing no nicotine.
- JUUL + No Patch: Participants were given Juul e-cigarettes for four weeks; in Switch Week 1 - half of participants used active nicotine patches and half used placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 used placebo patches during Switch Week 2, and the participants who received placebo patches during Switch Week 1 used active nicotine patches during Switch Week 2. AEs were assessed during Switch Weeks as well as during times when participants were smoking as usual and/or using JUUL, but not using nicotine patches.
  These data are AEs for subjects during the weeks that they were using JUUL and No Patches.
  Juul Electronic cigarette: The Juul e-cigarette pods contain 0.7 ml nicotine by volume / 5% nicotine by weight.
- VLNC + Active Patch: Participants were given very low nicotine cigarettes (VLNCs) for four weeks; in Switch Week 1 - half of participants used active nicotine patches and half used placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 used placebo patches during Switch Week 2, and the participants who received placebo patches during Switch Week 1 used active nicotine patches during Switch Week 2. AEs were assessed during Switch Weeks as well as during times when participants were smoking as usual and/or using VLNC, but not using nicotine patches.
  These data are AEs for subjects during the weeks that they were using VLNCs and Active Patches.
  Very Low Nicotine Cigarettes: These very low nicotine cigarettes (VLNCs) consist of reduced nicotine cigarettes containing 0.03 mg of nicotine; these VLNCs were obtained from National Institute on Drug Abuse (NIDA's) Drug Supply Program (NOT-DA-14-004).
  Active Nicotine Patch: Active nicotine patches, with dosing based on the package insert (>10 cigs/day = 21 mg patch and <11 cigs/day = 14 mg patches).
- VLNC + Placebo Patch: Participants were given very low nicotine cigarettes (VLNCs) for four weeks; in Switch Week 1 - half of participants used active nicotine patches and half used placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 used placebo patches during Switch Week 2, and the participants who received placebo patches during Switch Week 1 used active nicotine patches during Switch Week 2. AEs were assessed during Switch Weeks as well as during times when participants were smoking as usual and/or using VLNC, but not using nicotine patches.
  These data are AEs for subjects during the week that they were using VLNCs and Placebo Patches.
  Very Low Nicotine Cigarettes: These very low nicotine cigarettes (VLNCs) consist of reduced nicotine cigarettes containing 0.03 mg of nicotine; these VLNCs were obtained from National Institute on Drug Abuse (NIDA's) Drug Supply Program (NOT-DA-14-004).
  Placebo Patch: Placebo patch containing no nicotine.
- VLNC + No Patch: Participants were given very low nicotine cigarettes (VLNCs) for four weeks; in Switch Week 1 - half of participants used active nicotine patches and half used placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 used placebo patches during Switch Week 2, and the participants who received placebo patches during Switch Week 1 used active nicotine patches during Switch Week 2. AEs were assessed during Switch Weeks as well as during times when participants were smoking as usual and/or using VLNC, but not using nicotine patches.
  These data are AEs for subjects during the week that they were using VLNC and No Patches.
  Very Low Nicotine Cigarettes: These very low nicotine cigarettes (VLNCs) consist of reduced nicotine cigarettes containing 0.03 mg of nicotine; these VLNCs were obtained from National Institute on Drug Abuse (NIDA's) Drug Supply Program (NOT-DA-14-004).
- No Product + Active Patch: Participants were given no alternative nicotine delivery products but in Switch Week 1 - half of participants used active nicotine patches and half used placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 used placebo patches during Switch Week 2, and the participants who received placebo patches during Switch Week 1 used active nicotine patches during Switch Week 2. AEs were assessed during Switch Weeks as well as during times when participants were smoking as usual but not using nicotine patches.
  These data are AEs for subjects during the week that they were using No Product and Active Patches.
  Active Nicotine Patch: Active nicotine patches, with dosing based on the package insert (>10 cigs/day = 21 mg patch and <11 cigs/day = 14 mg patches).
- No Product + Placebo Patch: Participants were given no alternative nicotine delivery products but in Switch Week 1 - half of participants used active nicotine patches and half used placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 used placebo patches during Switch Week 2, and the participants who received placebo patches during Switch Week 1 used active nicotine patches during Switch Week 2. AEs were assessed during Switch Weeks as well as during times when participants were smoking as usual but not using nicotine patches.
  These data are AEs for subjects during the week that they were using No Product and Placebo Patches.
  Placebo Patch: Placebo patch containing no nicotine.
- No Product + No Patch: Participants were given no alternative nicotine delivery products but in Switch Week 1 - half of participants used active nicotine patches and half used placebo patches, in Switch Week 2 - the participants who received active nicotine patches during Switch Week 1 used placebo patches during Switch Week 2, and the participants who received placebo patches during Switch Week 1 used active nicotine patches during Switch Week 2. AEs were assessed during Switch Weeks as well as during times when participants were smoking as usual but not using nicotine patches.
  These data are AEs for subjects during the week that they were using No Product and No Patches.
Arm/Group | JUUL + Active Patch | JUUL + Placebo Patch | JUUL + No Patch | VLNC + Active Patch | VLNC + Placebo Patch | VLNC + No Patch | No Product + Active Patch | No Product + Placebo Patch | No Product + No Patch
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54 | 0/54 | 0/53 | 0/53 | 0/53 | 0/53 | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54 | 0/54 | 0/53 | 0/53 | 0/53 | 0/53 | 0/53 | 2/53
Other Adverse Events (participants affected / at risk) | 31/54 | 19/54 | 34/54 | 21/53 | 12/53 | 15/53 | 16/53 | 7/53 | 8/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JUUL + Active Patch (N=54) | JUUL + Placebo Patch (N=54) | JUUL + No Patch (N=54) | VLNC + Active Patch (N=53) | VLNC + Placebo Patch (N=53) | VLNC + No Patch (N=53) | No Product + Active Patch (N=53) | No Product + Placebo Patch (N=53) | No Product + No Patch (N=53)
Ruptured Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stroke (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JUUL + Active Patch (N=54) | JUUL + Placebo Patch (N=54) | JUUL + No Patch (N=54) | VLNC + Active Patch (N=53) | VLNC + Placebo Patch (N=53) | VLNC + No Patch (N=53) | No Product + Active Patch (N=53) | No Product + Placebo Patch (N=53) | No Product + No Patch (N=53)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Itching or Hives (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Skin Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 1 (2) | 2 (2) | 2 (2)
Insomnia (Nervous system disorders) | 4 (4) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Vivid Dreams (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weakness (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irregular Heartbeat (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trouble Breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 5 (6) | 9 (12) | 4 (5) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever/Chills (General disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling in face or hands (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 4 (4) | 3 (3) | 3 (3) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT04084210/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT04084210/ICF_001.pdf